CLINICAL TRIAL: NCT01028794
Title: Phase 1/2A Study of Intravenous Autologous Bone Marrow Mononuclear Cell Transplantation for Patients After Cerebral Embolism
Brief Title: Autologous Bone Marrow Mononuclear Cell Transplantation for Stroke Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Institute of Biomedical Research and Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Akihiko Taguchi, guest investigator, National Cerebral and Cardiovascular Center, Japan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000001133; UMIN000001133 (Other: University hospital Medical Information Network in Japan)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Cerebral Embolism; Stroke
Keywords: stroke; bone marrow; mononuclear cell; angiogenesis; neurogenesis
MeSH Terms: conditions — Intracranial Embolism; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- autologous bone marrow mononuclear cell (Experimental): On day 7-10 after stroke, patient has 25ml of bone marrow cells aspiration. Mononuclear cells are purified by Ficoll and administrated intravenously.
  Interventions: Biological: autologous bone marrow mononuclear cells
- autologous bone marrow mononuclear cells (Experimental): On day 7-10 after stroke, patient has 50ml of bone marrow cells aspiration. Mononuclear cells are purified by Ficoll and administrated intravenously.
  Interventions: Biological: autologous bone marrow mononuclear cells

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cells — intravenous administration of autologous bone marrow derived mononuclear cells obtained from 25ml of bone marrow on day 7-10 after stroke (only once in that period)
  Arms: autologous bone marrow mononuclear cell
Biological: autologous bone marrow mononuclear cells — intravenous administration of autologous bone marrow derived mononuclear cells obtained from 50ml of bone marrow on day 7-10 after stroke (only once in that period)
  Arms: autologous bone marrow mononuclear cells

SUMMARY:
The purpose of this study is to determine whether autologous bone marrow mononuclear cells transplantation after stroke is safe and/or effective to improve neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebral embolism.
* NIHSS score is more than (or equal to) 10.
* On day 7 after onset of stroke, the improvement of NIHSS is less than (or equal to) 5, compared with the level at administration.
* Bone marrow aspiration can be done in 10 days after onset of stroke

Exclusion Criteria:

* Patient with cerebral hemorrhage or symptomatic hemorrhagic infarction.
* Patient who expects brain surgery.
* Patient with acute myocardial infarction.
* Patient with coagulation disorder.
* Number of Platelet < 100000/mm3
* Serum creatinine level >2.0mg/dl
* Patient with malignancy.
* Patient with uncontrolled proliferative diabetic retinopathy.
* Patient suspected infective endocarditis.
* HBV, HCV, HIV or HTLV positive

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Improvement of NIHSS（National Institute of Health Stroke Scale） | 30 days after treatment
Frequency of change for the worse in NIHSS | 30 days aftrer treatment

SECONDARY OUTCOMES:
Mean level of mRS (modified Rankin Scale) | 30 days after treatment
Frequency of death | day 30 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko Taguchi, MD.PhD, Principal Investigator — Department of Cerebrovascular Disease, National Cardiovascular Center
Locations (1):
- Department of Cerebrovascular Disease, National Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Background] Taguchi A, Soma T, Tanaka H, Kanda T, Nishimura H, Yoshikawa H, Tsukamoto Y, Iso H, Fujimori Y, Stern DM, Naritomi H, Matsuyama T. Administration of CD34+ cells after stroke enhances neurogenesis via angiogenesis in a mouse model. J Clin Invest. 2004 Aug;114(3):330-8. doi: 10.1172/JCI20622. PMID 15286799
- [Background] Taguchi A, Ohtani M, Soma T, Watanabe M, Kinosita N. Therapeutic angiogenesis by autologous bone-marrow transplantation in a general hospital setting. Eur J Vasc Endovasc Surg. 2003 Mar;25(3):276-8. doi: 10.1053/ejvs.2002.1831. No abstract available. PMID 12623341
- [Background] Taguchi A, Matsuyama T, Moriwaki H, Hayashi T, Hayashida K, Nagatsuka K, Todo K, Mori K, Stern DM, Soma T, Naritomi H. Circulating CD34-positive cells provide an index of cerebrovascular function. Circulation. 2004 Jun 22;109(24):2972-5. doi: 10.1161/01.CIR.0000133311.25587.DE. Epub 2004 Jun 7. PMID 15184275
- [Background] Taguchi A, Wen Z, Myojin K, Yoshihara T, Nakagomi T, Nakayama D, Tanaka H, Soma T, Stern DM, Naritomi H, Matsuyama T. Granulocyte colony-stimulating factor has a negative effect on stroke outcome in a murine model. Eur J Neurosci. 2007 Jul;26(1):126-33. doi: 10.1111/j.1460-9568.2007.05640.x. PMID 17614944